

## INTEGRATING HEPATOLOGICAL, NUTRITIONAL, AND COGNITIVE BEHAVIORAL THERAPY-BASED PSYCHOLOGICAL SUPPORT IS AN EFFECTIVE MULTIDISCIPLINARY APPROACH TO IMPROVE LONG-TERM CLINICAL OUTCOMES IN THE MANAGEMENT OF MASLD PATIENTS: A RANDOMIZED CLINICAL TRIAL [THE "COCONUT" STUDY]

Informed consent form

Version approved, 31 May 2023



## Azienda Ospedaliera Universitaria Università degli Studi della Campania "L. Vanvitelli" DAI di CHIRURGIA, ORTOPEDIA ED EPATOGASTROENTEROLOGIA

## UNITA' OPERATIVA COMPLESSA DI EPATO-GASTROENTEROLOGIA

## **INFORMED CONSENT FORM FOR THE STUDY**

| Brief title of th | ne study | Integrating hepatological, nutritional, and psychological support as a multidisciplinary management to improve long-term clinical outcomes in MASLD |
|---|---|---|
| ACRONYM | | CoCoNut |
| The undersigned | | <b>,</b> |
| Born on | to | resident in |
| I have received a | copy of the study informat | oroviding any reason and without this impacting my usual healthcare. Sion, the informed consent form, the privacy policy, and the consentinals are kept at the center. |
| | · | articipate in the above-mentioned study, therefore: |
| l consent to | the processing of my de | mographic, clinical, anthropometric and therapeutic data |
| Date | Patient's signature | |
| Date | Signature of the doctor who | nformed the patient |
| Date | Signature of the participant's (only in case of patient inabili | legal representative/guardian |